CLINICAL TRIAL: NCT05326308
Title: Zanubrutinib (Brukinsa®) in Patients With Waldenström's Macroglobulinemia (WM), Chronic Lymphocytic Leukemia (CLL), Marginal Zone Lymphoma (MZL) and Follicular Lymphoma (FL) - a Prospective Multicenter Observational Cohort Study
Brief Title: Zanubrutinib in Patients With Waldenström's Macroglobulinemia, Chronic Lymphocytic Leukemia, Marginal Zone Lymphoma and Follicular Lymphoma
Acronym: ARIADNE
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: BeOne Medicines I GmbH Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOM-100461
Record Dates: First submitted 2022-03-23; First posted 2022-04-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Waldenström's Macroglobulinemia; Chronic Lymphocytic Leukemia; Marginal Zone Lymphoma; Follicular Lymphoma
Keywords: Waldenström's Macroglobulinemia; Zanubrutinib; Brukinsa; Chronic Lymphocytic Leukemia; Marginal Zone Lymphoma; Follicular Lymphoma
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular | interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All patients will be asked to give additional informed consent that their routinely collected biomaterial will be assigned to the decentralized biobank and may be used for future translational research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Waldenström's Macroglobulinemia: 75 patients (excluding screening failures, patients with off-label use or with violation of inclusion/exclusion criteria identified after treatment start) receiving zanubrutinib (Brukinsa®)
  Interventions: Drug: Zanubrutinib
- Chronic Lymphocytic Leukemia: 450 patients (excluding screening failures, patients with off-label use or with violation of inclusion/exclusion criteria identified after treatment start) receiving zanubrutinib (Brukinsa®)
  Interventions: Drug: Zanubrutinib
- Marginal Zone Lymphoma: 40 patients (excluding screening failures, patients with off-label use or with violation of inclusion/exclusion criteria identified after treatment start) receiving zanubrutinib (Brukinsa®)
  Interventions: Drug: Zanubrutinib
- Follicular Lymphoma: 40 patients (excluding screening failures, patients with off-label use or with violation of inclusion/exclusion criteria identified after treatment start) receiving zanubrutinib (Brukinsa®) in combination with obinutuzumab (Gazyvaro®)
  Interventions: Drug: Zanubrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib — according to the Summary of Product Characteristics (SmPC).
  Other Names: Brukinsa®
Drug: Obinutuzumab — according to the Summary of Product Characteristics (SmPC).
  Other Names: Gazyvaro®
  Groups: Follicular Lymphoma

SUMMARY:
The objective of this NIS is to evaluate medical resource utilization, where data is rare in all cohorts, patient's QoL and effectiveness of zanubrutinib treatment in adult patients with WM, CLL, MZL and FL in a real-world setting.

DETAILED DESCRIPTION:
ARIADNE will collect and analyze data of adult patients with WM, CLL, MZL or FL in need of treatment. The study will explore the medical resource utilization during therapy with zanubrutinib (Brukinsa®). Further aims are to assess effectiveness, safety and tolerability of the treatment as well as treatment satisfaction and biomarkers. These data will be supplemented by the assessment of patient-reported outcomes (PROs)/ health-related quality of life (QoL).

Since treatment options for MW, CLL, MZL or FL are limited and the most important factor is to keep or improve QoL of the patients, there is an urge for real-world clinical data of patients treated with zanubrutinib, especially focusing on patients already treated upfront with a BTK inhibitor, older patients and patients with comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Waldenström's macroglobulinemia (all treatment lines) OR
* Chronic lymphocytic leukemia (all treatment lines) OR
* Marginal zone lymphoma (≥2 treatment line and at least one anti-CD20 antibody-based previous therapy)
* Follicular lymphoma (≥3 treatment line)
* Signed and dated informed consent form
* Treatment with zanubrutinib according to current SmPC for WM, CLL and MZL
* Treatment with zanubrutinib + obinutuzumab for FL according to current SmPC
* Treatment decision before inclusion into this non-interventional study
* Age ≥18 years.

Exclusion Criteria:

* Contraindications according to SmPC for patients with WM, CLL, MZL or FL
* Participation in an interventional clinical trial during zanubrutinib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Waldenström's macroglobulinemia (WM), Chronic Lymphocytic Leukemia (CLL), Marginal Zone Lymphoma (MZL) or Follicular Lymphoma (FL) in need of treatment with decision for treatment with zanubrutinib (Brukinsa®) according to the Summary of Product Characteristics (SmPC).
Sampling Method: Non-Probability Sample
Enrollment: 705 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Medical resource utilization | During zanubrutinib treatment, up to 6.3 years
  Frequency of hospitalizations, i.e. number of hospital stays plus number of emergency unit visits (without hospitalization) per patient

SECONDARY OUTCOMES:
Global health-related quality of life (QoL) collected via EORTC QLQ-C30 during course of treatment and follow-up | During zanubrutinib treatment and follow-up, up to 6.3 years
  Course of QoL during treatment and follow-up (collected via European Organisation for research and treatment of cancer quality of life in cancer patient questionnaire (EORTC QLQ-C30). Scoring of the questionnaire will be performed according to the respective manual.
Global health-related quality of life (QoL) collected via EQ-5D-5L during course of treatment and follow-up | During zanubrutinib treatment and follow-up, up to 6.3 years
  Course of QoL during treatment and follow-up (collected via European quality of life 5 dimension 5 level version (EQ-5D-5L)). Scoring of the questionnaire will be performed according to the respective manual.
Incidence of (serious) adverse events ((S)AEs) | Start of zanubrutinib treatment until 30 days after end of zanubrutinib treatment
  Incidence of (S)AEs; (S)AEs will be summarized by the most recent Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term.
Incidence of (serious) adverse drug reactions ((S)ADRs) | Start of zanubrutinib treatment until end of study, up to 6.3 years
  Incidence of (S)ADRs related to zanubrutinib
Incidence of adverse events of special interest (AESIs) | Start of zanubrutinib treatment until 30 days after end of zanubrutinib treatment
  Incidence of AESIs
Time to AESIs | Start of zanubrutinib treatment until 30 days after end of zanubrutinib treatment
  The time to first onset of AESIs.
Time to neutropenia | Start of zanubrutinib treatment until 30 days after end of zanubrutinib treatment
  The time to first onset of neutropenia grade ≥3 (MedDRA terms: neutropenia and neutrophil count decrease).
Rate of neutropenia grade ≥3 | Start of zanubrutinib treatment until 30 days after end of zanubrutinib treatment
  Rate of patients with neutropenia grade ≥3 during zanubrutinib treatment. Neutropenia incorporates the MedDRA terms: neutropenia and neutrophil count decrease.
Proportion of patients with complete response (CR) or very good partial response (VGPR) (best reported response) | During zanubrutinib treatment, up to 6.3 years
  The proportion of patients with a best overall response of CR or VGPR.
In the WM cohort only: Major response rate (MRR) | During zanubrutinib treatment, up to 6.3 years
  MRR is defined as the proportion of patients with a best overall response ≥ PR (partial response)
In the WM cohort only: Best response | During zanubrutinib treatment, up to 6.3 years
  Best response is defined as best reported response during study treatment CR (complete response) or VGPR (very good partial response).
In the WM cohort only: IgM levels | During zanubrutinib treatment, up to 6.3 years
  Change of IgM levels until end of zanubrutinib treatment for WM cohort.
Progression-free Survival (PFS) | Treatment start with zanubrutinib until end of study, up to 6.3 years
  PFS is defined as the time from treatment start until progression or death from any cause, whichever comes first.
6-, 12-, 18- and 24-month PFS rate | 6, 12, and 24 months after start of zanubrutinib treatment
  Percentage of patients without disease progression or death from any cause at 6, 12, and 24 months after start of zanubrutinib treatment.
Overall Survival (OS) | Treatment start with zanubrutinib until end of study, up to 6.3 years
  OS is defined as the time from treatment start until death.
6-, 12-, 18- and 24-month OS rate | 6, 12, and 24 months after start of zanubrutinib treatment
  Percentage of patients alive at 6, 12, and 24 months after start of zanubrutinib treatment.
WM Cohort: Overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the WM cohort, overall response rate is defined as CR, VGPR and PR (partial response).
WM Cohort: Best overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the WM cohort, best overall response rate is defined as CR, VGPR, PR (partial response), MR (minor response), SD (stable disease) or PD (progressive disease).
CLL Cohort: Overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the CLL cohort, overall response rate is defined as CR and PR.
CLL Cohort: Best overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the CLL cohort, best overall response rate is defined as CR, PR, SD or PD.
MZL Cohort: Overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the MZL cohort, overall response rate is defined as CR, pMRD (probable minimal residue disease), PR and rRD (responding residual disease).
MZL Cohort: Best overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the MZL cohort, best overall response rate is defined as CR, pMRD, PR, rRD, No change/SD or PD
FL Cohort: Overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the FL cohort, overall response rate is defined as CR or PR.
FL Cohort: Best overall response rate (ORR) | During zanubrutinib treatment, up to 6.3 years
  For the FL cohort, best overall response rate is defined as CR, PR, MR, SD or PD.
Time to treatment failure (TTF) | Treatment start with zanubrutinib until end of treatment, up to 6.3 years
  TTF is defined as time interval from treatment start to discontinuation of treatment because of disease progression, treatment toxicity, switch of therapy of any reason, and death.
Frequency of blood product transfusion | During zanubrutinib treatment, up to 6.3 years
  The number of patients receiving blood product transfusion, the number of transfusions per patient and the kind of transfusion (e.g., erythrocytes, thrombocytes).
WM Cohort: Change of IgM levels until end of zanubrutinib treatment | Baseline and end of zanubrutinib treatment, up to 6.3 years
  Difference between the baseline value and the end of treatment value of the IgM level.
Therapy decision making | Baseline
  Frequency and weighting of distinct parameters affecting therapy choice of the treating physician assessed by project specific questionnaire
Time from first diagnosis of WM, CLL, MZL or FL to zanubrutinib treatment start | Baseline
  Time from first diagnosis of WM, CLL, MZL or FL to zanubrutinib treatment start including timing and duration of possible watch & wait strategy.
Previous therapies | Baseline
  Key details of previous therapies (including plasmapheresis for WM, transplantations for WM, CLL and FL, radiotherapy for CLL, MZL and FL and surgery for CLL, MZL and FL).
Daily dose of zanubrutinib | During zanubrutinib treatment, up to 6.3 years
  Frequency tables including the daily dose (mg) will be given using descriptive statistics.
FL cohort: Daily dose of obinutuzumab | During zanubrutinib treatment, up to 6.3 years
  Frequency tables including the daily dose (mg) will be given using descriptive statistics.
Dose modifications of zanubrutinib | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including therapy modifications (reduction and increase) with reasons using descriptive statistics.
FL cohort: Dose modifications of obinutuzumab | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including therapy modifications (reduction and increase) with reasons using descriptive statistics.
Therapy interruptions of zanubrutinib | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including treatment interruptions with reasons as well as reasons for treatment termination.
FL cohort: Therapy interruptions of obinutuzumab | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including treatment interruptions with reasons as well as reasons for treatment termination.
Dose intensity of zanubrutinib | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including the dose intensity (absolute and relative) using descriptive statistics.
FL cohort: Dose intensity of obinutuzumab | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including the dose intensity (absolute and relative) using descriptive statistics.
Treatment duration with zanubrutinib | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including the treatment duration will be given using descriptive statistics.
FL cohort: Treatment duration with obinutuzumab | During zanubrutinib treatment, up to 6.3 years
  Frequency tables will be provided including the treatment duration will be given using descriptive statistics.
Subsequent antineoplastic therapies | End of zanubrutinib treatment until end of study, up to 6.3 years
  Key details of subsequent antineoplastic therapies after zanubrutinib (including plasmapheresis for WM, stem cell transplantations for WM, CLL and FL, radiotherapy for CLL, MZL and FL and surgery for CLL, MZL and FL): duration (descriptive statistics), number, substances and reason for end of subsequent treatments (frequencies).
Frequency for concomitant medication during zanubrutinib treatment | During zanubrutinib treatment, up to 6.3 years
  Substances (WHO-ATC level 2), ongoing status and indication (frequencies)
Frequency of antibiotic use for prophylactic reasons during zanubrutinib treatment | During zanubrutinib treatment, up to 6.3 years
  Proportion of patients with at least one-time antibiotic use for prophylactic reasons during zanubrutinib treatment.
Frequency of antibiotic use for treatment of AEs during zanubrutinib treatment | During zanubrutinib treatment, up to 6.3 years
  Proportion of patients taking at least one-time antibiotics for treatment of AEs during zanubrutinib treatment.
Frequency of antibiotic use in patients with neutropenia during zanubrutinib treatment | During zanubrutinib treatment, up to 6.3 years
  Proportion of patients presenting with neutropenia during zanubrutinib treatment taking at least one-time antibiotics.

OTHER OUTCOMES:
Patients' treatment expectation and satisfaction | Baseline, 3 months after treatment start with zanubrutinib, end of treatment
  Patients' treatment expectation and satisfaction (assessed via project specific questionnaire) will be analyzed by time point, using absolute and relative frequencies.
Physicians' treatment expectation and satisfaction | Baseline, 3 months after treatment start with zanubrutinib, end of treatment
  Physicians' treatment expectation and satisfaction (assessed via project specific questionnaire) will be analyzed by time point, using absolute and relative frequencies.
Collection of biomarker test results (according to clinical routine) | Baseline, up to 6.3 years
  Number of patients with biomarker testing as well as sample types, test methods and test results of biomarker testing per biomarker will be provided including patients with resistance mechanism testing before treatment decision with zanubrutinib. Information on the testing of MYD88 and CXCR4 is mandatory.
Patient management during SARS-Covid-19 pandemic | Baseline and end of zanubrutnib treatment, up to 6.3 years
  The patient management during SARS-Covid-19 pandemic (assessed via project specific questionnaire) (patient supervised by oncologist or additionally by family doctor) will be presented by frequency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kisro, Dr., Principal Investigator — Lübecker Onkologische Schwerpunktpraxis; Richard Greil, Prof., Principal Investigator — Universitätsklinikum Salzburg, Klinik für Innere Medizin III
Locations (2):
- Universitätsklinikum Salzburg, Klinik für Innere Medizin III, Salzburg, Austria
- Lübecker Onkologische Schwerpunktpraxis, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No